CLINICAL TRIAL: NCT02904018
Title: Validation Study of Oral Teleconsultation - Study EDENT2
Brief Title: Validation Study of Oral Teleconsultation
Acronym: EDENT2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9370
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2014-02

CONDITIONS: Dental Care
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: teleconsultation — Patients performing oral care required as a result of their diagnosis by teleconsultation in vulnerable populations (elderly, disabled adults).

SUMMARY:
In this study we want to evaluate the oral care pathway after an oral teleconsultation.

DETAILED DESCRIPTION:
An oral teleconsultation was proposed to the 461 residents of the public hospital of Uzès. A specifically trained nurse recorded 4 videos (1 per quadrant) per mouth with an intra-oral camera using fluorescent light (Soprocare®) and keyed in information about the resident (general state, identification,…). These data were recorded and sent onto a central secured server, through a specific piece of software (e-DENT®). The dentists from the University Hospital of Montpellier were then able to analyse the videos remotely, make a diagnosis and organise each resident's oral care.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged at least 18 years
* Patients cared for in their host institution

Exclusion Criteria:

* NA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are in long-term care home with oral telemedicine activity
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic of caries | 1 day
  Teleconsultation will be made using a specific camera SoproCare®6, the company Acteon

SECONDARY OUTCOMES:
Diagnostic of caries | 6 months
  Teleconsultation will be made using a specific camera SoproCare®6, the company Acteon

IPD SHARING:
Plan to Share IPD: Undecided